CLINICAL TRIAL: NCT01405352
Title: The Effect of Vitamin A Supplementation on CD4+ T-cell Secretion in Obese Individuals
Brief Title: The Effect of Vitamin A Supplementation on Cytokine Profile in Obesity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Ali Akbar Saboor Yaraghi/Assistant professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 89-04-27-11869
Record Dates: First submitted 2011-02-14; First posted 2011-07-29 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Obesity
Keywords: obesity; vitamin A; immune system
MeSH Terms: conditions — Obesity | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Non obese/ vitamin A (Active Comparator): Non obese individuals with body mass index 18.5-24.9 kg/m2 who receive 25000 IU/day vitamin A for 4 months .
  Interventions: Dietary Supplement: Vitamin A
- obese/ placebo (Placebo Comparator): obese individuals with body mass index greator than 30 kg/m2 who receive 1 cap placebo per day for 4 months .
  Interventions: Dietary Supplement: Vitamin A
- Obese/ vitamin A (Active Comparator): obese individuals with body mass index greater than 30 kg/m2 who receive 25000 IU/day vitamin A for 4 months
  Interventions: Dietary Supplement: Vitamin A

INTERVENTIONS:
Dietary Supplement: Vitamin A — 25000 IU/day vitamin A 4 months
  1 Cap/Day
  1 cap placebo/day for 4 month

SUMMARY:
In this double blind placebo controlled trial,cytokine secretion of CD4+ T-cells after 4 month supplementation of vitamin A will be compared with placebo intaking group.

DETAILED DESCRIPTION:
Obesity is a chronic disease consisting of the increase in body fat stores. Obesity is an important health concern because of its well known relationships with metabolic and endocrine disorders such as cardiovascular disease, type 2 diabetes, hypertension and immune dysfunction. Low-grade systemic inflammation, confirmed by the increase of inflammatory markers such as C-reactive protein and interleukin-6 has been observed in obesity. CD4+ T-helpers are the most important regulators of immune system. Epidemiological evidence has linked obesity to several (but not all) autoimmune disorders, including inflammatory bowel disease (IBD) and psoriasis .Some sublineages of T- helpers plays core roles in immune dysfunction, and recent evidence demonstrates that an imbalance of T-cell subgroups including Th1, Th2, Th17 and Treg has occurred in obesity. This imbalance is the redirection of the immune response from most often Th2 and Treg like responses to Th1 and Th17 like responses respectively, however the opposite is desired. Vitamin A (VA) or VA-like analogs known as retinoids, are potent hormonal modifiers of type 1 or type 2 responses but a definitive description of their mechanism(s) of action is lacking. High level dietary vitamin A enhances Th2 cytokine production and IgA responses, and is likely to decrease Th1 cytokine production. Retinoic acid inhibits IL-12 production in activated macrophages, and RA pretreatment of macrophages reduces IFNγ and TNF α production and increases IL4 production in antigen primed CD4 T cells. Supplemental treatment with vitamin A or retinoic acid (RA) decreases IFNγ and increases IL5, IL10, and IL4 production.

ELIGIBILITY:
Inclusion Criteria:

waist to hip ratio >0.8 and BMI>30 kg/m2 for obese individuals waist to hip ratio <0.8 and BMI 18.5 - 24.9 kg/m2 for Non obese individuals

Exclusion Criteria:

* subjects who have diseases which affect on Th1/Th2 balance such as asthma, active viral infections, and autoimmune diseases, OR
* subjects with pregnancy, lactation, menopause, diabetes
* subjects who have allergy to vitamin A compounds, OR
* subjects who have used vitamin supplements or in last 3 months, OR
* subjects with morbid obesity(BMI >40 kg/m2),OR
* overweight subjects (25 <BMI<29.9 kg/m2)

Ages: 20 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Complete Blood Count-diff | Change from baseline at 4 months
Serum HDL concentrations | Change from baseline at 4 months
Serum LDL concentrations | Change from baseline at 4 months
Serum total cholesterol concentrations | Change from baseline at 4 months
Serum Triglycerides concentrations | Change from baseline at 4 months
Serum SGOT concentrations | Change from baseline at 4 months
Serum SGPT concentrations | Change from baseline at 4 months
Serum T3 concentrations | Change from baseline at 4 months
Serum T4 concentrations | Change from baseline at 4 months
Serum TSH concentrations | Change from baseline at 4 months
Serum FBS concentrations | Change from baseline at 4 months
Serum CRP concentrations | Change from baseline at 4 months
Serum RF concentrations | Change from baseline at 4 months

SECONDARY OUTCOMES:
Serum IL-2 concentrations | Change from baseline at 4 months
Serum IL-6 concentrations | Change from baseline at 4 months
Serum IL-10 concentrations | Change from baseline at 4 months
Serum IL-12 concentrations | Change from baseline at 4 months
Serum IL-13 concentrations | Change from baseline at 4 months
Serum IL-17 concentrations | Change from baseline at 4 months
Seum IL-1β concentrations | Change from baseline at 4 months
Serum TGF β concentrations | Change from baseline at 4 months
serum IFN γ concentrations | Change from baseline at 4 months
serum Angiotensin П concentrations | Change from baseline at 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences, School of Public Health, Tehran, Tehran Province, Iran